CLINICAL TRIAL: NCT02287662
Title: The Vancouver Multidisciplinary, Multimodality, But Minimalist Clinical Pathway Facilitates Safe Next Day Discharge Home at Low, Medium, and High Volume Transfemoral Transcatheter Aortic Valve Replacement Centres: The 3M TAVR Study
Brief Title: The Multidisciplinary, Multimodality, But Minimalist Approach to Transfemoral Transcatheter Aortic Valve Replacement
Acronym: 3MTAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BC Centre for Improved Cardiovascular Health (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vancouver 3M Clinical Pathway (Experimental): The Vancouver 3M Clinical Pathway utilizes objective anatomical and functional screening criteria as well as strict peri-procedural guidelines to determine if next day discharge home is appropriate.
  Interventions: Other: Vancouver 3M Clinical Pathway

INTERVENTIONS:
Other: Vancouver 3M Clinical Pathway

SUMMARY:
The primary objective of this study is to determine the efficacy, safety and feasibility of next day discharge home in patients undergoing balloon-expandable transfemoral TAVR utilizing the Vancouver 3M Clinical Pathway in low, medium, and high volume North American centres.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe symptomatic aortic stenosis undergoing elective transfemoral TAVR with a balloon expandable transcatheter heart valve

1. Considered at increased surgical risk by the Multidisciplinary Heart Team.
2. Informed written consent

Exclusion Criteria:

1. Non -cardiovascular co-morbidity reducing life expectancy to < 3 years
2. Any factor precluding 1 year follow-up
3. Inadequate CT image acquisition to perform area-based annular CT sizing, exclude adverse root features, and determine a coaxial valve deployment angle (CT is not required for valve-in-valve procedures)
4. Predicted inability to perform uncomplicated percutaneous vascular access and closure
5. Iliofemoral diameter < 6 mm for SAPIEN XT or <5.5 mm for SAPIEN 3 (measured at or above the mid-femoral head)
6. Inpatient (unless clinically stable, mobilizing at baseline, and primarily in hospital for logistical reasons.
7. Significant communication barrier(s) that interfere with ability to follow peri-procedural and discharge instructions
8. MMSE < 24/30 (unless language barrier or limited formal education), 5-metre gait > 7 seconds (unless chronic mobility impairment not affecting ability to perform ADLs), and ADL < 6/6
9. Insufficient social support to facilitate next day discharge
10. Airway unfavourable for emergent intubation
11. Inability to lay supine without conscious sedation or general anesthetic
12. Not receiving a balloon expandable transcatheter heart valve

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 411 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The composite of all-cause mortality or stroke | 30 days post-procedure
The proportion of patients undergoing elective transfemoral TAVR using the Vancouver 3M Clinical Pathway, who are discharged the next day | Next day

SECONDARY OUTCOMES:
All-cause mortality | 30 days post-procedure
Stroke | 30 days post-procedure
30-day major vascular complications | 30 days post-procedure
30-day major/life-threatening bleed | 30 days post-procedure
Any readmission to hospital within 30 days | 30 days post-procedure
> mild paravalvular regurgitation | Post-procedure/discharge
New permanent pacemaker | 30 days post-procedure
Conversion to general anesthetic/intubation | Peri-procedure
Myocardial infarction | Peri-procedure
Repeat procedure for valve-related dysfunction | 30 days post-procedure
Stage 3 acute kidney injury (need for dialysis) | 30 days post-procedure
Patient-centred outcomes including health related quality of life as measured by KCCQ and SF-12 at baseline, 2 weeks, 30 days, and 1 year | Baseline, and 2 weeks, 30 day and 1 year post procedure
Economic evaluation including health resource utilization, and cost effectiveness | Peri- and post-procedure
Death or stroke at one year | 1 year post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: David A Wood, MD, Principal Investigator — University of British Columbia; John A Webb, MD, Principal Investigator — University of British Columbia
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Butala NM, Wood DA, Li H, Chinnakondepalli K, Lauck SB, Sathananthan J, Cairns JA, Magnuson EA, Barker M, Webb JG, Welsh R, Cheung A, Ye J, Velianou JL, Wijeysundera HC, Asgar A, Kodali S, Thourani VH, Cohen DJ; 3M-TAVR Investigators. Economics of Minimalist Transcatheter Aortic Valve Replacement: Results From the 3M-TAVR Economic Study. Circ Cardiovasc Interv. 2022 Oct;15(10):e012168. doi: 10.1161/CIRCINTERVENTIONS.122.012168. Epub 2022 Oct 18. PMID 36256698